CLINICAL TRIAL: NCT05340374
Title: Cabazitaxel in Combination With 177Lu-PSMA-617 in Metastatic Castration-resistant Prostate Cancer
Acronym: LuCAB
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21/018
Record Dates: First submitted 2022-04-14; First posted 2022-04-22 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; mCRPC
MeSH Terms: interventions — cabazitaxel; Pluvicto

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): In this single-arm study, patients will receive 7.4 GBq of 177Lu-PSMA-617 on Day 1 of every 6 week Cycle. Cabazitaxel will be administered concurrently on Day 2 and Day 23 of each Cycle (every 3 weeks). The dose of cabazitaxel will vary in dose-escalation. Up to 6 Cycles will be given.
  Interventions: Drug: Cabazitaxel; Drug: 177Lu-PSMA-617

INTERVENTIONS:
Drug: Cabazitaxel — Cabazitaxel belongs to the Taxane group of drugs which function by interfering with microtubule depolymerisation and thus inhibit mitosis, which leads to cell death via apoptosis. It is the first chemotherapy agent to improve survival in patients with mCRPC with progressive disease after docetaxel-based treatment.
Drug: 177Lu-PSMA-617 — Lutetium-177 (177Lu)-PSMA is a radiopharmaceutical comprised of a small molecule inhibitor of PSMA that binds with high affinity to PSMA which is expressed on the prostate cancer cell, labelled with 177Lu. 177Lu has favourable characteristics for radionuclide therapy emitting both a short-range (1-2mm) cytotoxic beta-particle, minimising irradiation of non-targeted normal tissues, alongside gamma emission that allows imaging. Multiple clinical trials have demonstrated high clinical activity and limited normal tissue toxicity using 177Lu-PSMA-617.

SUMMARY:
This clinical trial will evaluate the safety of Cabazitaxel in combination with 177Lu-PSMA-617 in metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
This prospective, single-centre, single-arm, open label, phase I/II trial will assess the safety, efficacy and anti-tumour activity of cabazitaxel in combination with 177Lu-PSMA-617 in patients with metastatic castration-resistant prostate cancer (mCRPC).

This study aims to assess and establish the maximum tolerated dose (MTD), dose-limiting toxicities (DLTs), and recommended phase 2 dose (RP2D) of cabazitaxel in combination with 177Lu-PSMA-617 in patients with mCRPC.

32-44 men with mCRPC who have progressed on prior docetaxel and a second-generation AR antagonist will be enrolled in this trial in two stages: dose escalation and a dose expansion phase over a period of 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients aged 18 years or older at the time of informed consent.
2. Patient has provided written informed consent.
3. Histologically confirmed adenocarcinoma of the prostate without neuroendocrine or small cell differentiation.
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
5. Patients must have had prior treatment with docetaxel.
6. Patients must have progressed on a second-generation androgen receptor (AR)-targeted agent (e.g., enzalutamide, abiraterone, or apalutamide) in the castrate-resistant setting.
7. Patients must have progressive disease. The Prostate Cancer Clinical Trials Working Group 3 (PCWG3) defines this as any one of the following:

   1. PSA progression: minimum of two rising PSA values from a baseline measurement with an interval of ≥ 1 week between each measurement
   2. Soft tissue or visceral disease progression as per Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1) criteria
   3. Bone progression: ≥ 2 new lesions on bone scan
8. At least three weeks since the completion of surgery prior to registration.
9. Prior surgical orchiectomy or chemical castration maintained on luteinizing hormone-releasing hormone (LHRH) analogue (agonist or antagonist).
10. Serum testosterone levels ≤ 1.75nmol/L within 28 days prior to registration.
11. Imaging evidence of metastatic disease documented with either whole body bone scan (WBBS) or computed tomography (CT) scan performed within 28 days prior to registration.
12. Significant prostate-specific membrane antigen (PSMA) avidity on PSMA PET/CT, defined as a minimum uptake of SUVmax 15 at a site of disease.
13. Patients must have a life expectancy ≥ 12 weeks.
14. Assessed by a medical oncologist as suitable for treatment with cabazitaxel and 177Lu-PSMA-617.
15. Patients must have adequate bone marrow, hepatic and renal function documented within 28 days prior to registration, defined as:

    1. Haemoglobin ≥ 90 g/L independent of transfusions (no red blood cell transfusion in last 28 days prior to registration)
    2. Absolute neutrophil count (ANC) ≥ 1.5x10^9/L
    3. Platelets ≥ 150 x10^9/L
    4. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) except for patients with known Gilbert's syndrome, where this applies for the unconjugated bilirubin component
    5. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN if there is no evidence of liver metastasis or ≤ 5 x ULN in the presence of liver metastases
    6. Albumin ≥ 25 g/L
    7. Adequate renal function: patients must have a creatinine clearance estimated of ≥ 40 mL/min using the Cockcroft-Gault equation
16. Sexually active patients are willing to use medically acceptable forms of barrier contraception.
17. Willing and able to comply with all study requirements, including all treatments and the timing and nature of all required assessments.

Exclusion Criteria:

1. Superscan on WBBS or diffuse marrow disease on PSMA PET.
2. Site(s) of measurable disease that are FDG-positive with low PSMA expression (SUVmax <10).
3. Prior treatment with cabazitaxel or 177Lu-PSMA-617.
4. Contraindications to the use of corticosteroid treatment.
5. Other malignancies within the previous 2-years other than basal cell or squamous cell carcinomas of skin or other cancers that are unlikely to recur within 24 months.
6. Presence of untreated brain metastases or leptomeningeal metastases.
7. Patients with symptomatic or impending cord compression unless appropriately treated beforehand and clinically stable for ≥ four weeks.
8. Concurrent illness, including severe infection that may jeopardise the ability of the patient to undergo the procedures outlined in this protocol with reasonable safety.
9. Persistent toxicities (CTCAE v5.0 >/= Grade 2) caused by previous cancer therapy, excluding alopecia.
10. Known HIV or hepatitis B or C infection.
11. Radiotherapy or systemic anti-cancer therapies administered within 14 days prior to registration, excluding androgen deprivation therapy (ADT).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 35 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLTs) | Dose escalation phase is expected to be completed 9 months from the time the first patient is recruited.
  A DLT is defined as a toxicity that prevents further administration of the trial treatment at that dose level.
  Each cohort of 3 patients be assessed for DLTs in the first 6 weeks (cycle 1) of treatment and a dose for the next cohort will be determined.
Maximum Tolerated dose (MTD) | Dose escalation phase is expected to be completed 9 months from the time the first patient is recruited.
  The MTD is defined as the highest dose level at which the incidence of DLT was less than 2/6.
Recommended Phase 2 Dose (RP2D) | Up to 30 months from the time the first patient is recruited.
  After the MTD is established, additional patients will be treated at the MTD. Safety and efficacy data from the study will be used to define the RP2D.

SECONDARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) measured using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 | Through study completion, up until 24 months after the last patient commences treatment
  Safety of the combination will be measured by AEs and SAEs.
50% Prostate-Specific Antigen Response Rate (PSA-RR) | Through study completion, up until 24 months after the last patient commences treatment
  PSA will be assessed at baseline and every 3 weeks from cycle 1 day 1. PSA response will be defined as a 50% or greater decrease in PSA from baseline to the lowest post-baseline PSA result. A second consecutive value obtained 3 or more weeks later is required to confirm the PSA response.
Objective response rate (ORR) by Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST1.1) in patients with measurable disease | Through study completion, up until 24 months after the last patient commences treatment
  Objective Response (OR) is only applicable for the subset of patients with measurable disease by RECIST1.1. OR is defined as a partial response (PR) or complete response (CR) at any stage from time of commencement of protocol treatment to the time of subsequent systemic anti-cancer treatment. The ORR is calculated as the proportion of patients with a best response of CR or PR.
Radiographic Progression-Free Survival (rPFS) | Through study completion, up until 24 months after the last patient commences treatment
  rPFS is defined as the time from treatment initiation to the first date of documented radiographic progression using conventional imaging or death due to any cause, whichever occurs first. The radiographic progression will be assessed by the investigator per RECIST1.1 for soft tissue and Prostate Cancer Clinical Trials Working Group 3 (PCWG3) for bone lesions.
PSA progression free survival (PSA-PFS) | Through study completion, up until 24 months after the last patient commences treatment
  PSA-PFS is defined as the time from treatment initiation to the date of PSA progression per PCWG3 or death due to any cause, whichever occurs first. The date of PSA progression is the date that an increase of 25% or more and an absolute increase of 2ng/mL or more from the nadir is documented. For patients who have an initial PSA decline during treatment, this must be confirmed by a second value 3 or more weeks later.
Overall survival (OS) | Through study completion, up until 24 months after the last patient commences treatment
  OS is defined as the time from treatment initiation to the date of death due to any cause.
Describe pain within 12 months of treatment commencement | Through completion of 12 months after treatment commencement of last patient
  Pain will be assessed using the Brief Pain Inventory - Short Form (BPI-SF). This form assesses pain at its "worst," "least," "average," and "now" (current pain) in a 24-hour period at different timepoints, using a scale from 0-10. A higher score indicates more severe pain. The primary endpoint is the area under the curve (AUC) obtained from repeated patient responses to the BPI-SF item concerning "worst pain" in 24 hours.
  Pain will be assessed at baseline, 6 weeks, 3 months, 6 months, 9 months and 12 months and will be scored according to the respective manuals.
Describe health-related quality of life (QoL) within 12 months of treatment commencement | Through completion of 12 months after treatment commencement of last patient
  QoL will be assessed using the Functional Assessment of Cancer Therapy for Prostate Cancer (FACT-P) questionnaire. The primary endpoint for QoL is the area under the curve (AUC) of the trial outcome index (TOI), which is the sum of the Functional Assessment of Cancer Therapy -General (FACT-G), physical well-being, functional well-being, and prostate cancer subscale (PCS) scores. The score ranges from 0-156. A higher score indicates better quality of life.
  QoL will be assessed at baseline, 6 weeks, 3 months, 6 months, 9 months and 12 months and will be scored according to the respective manuals.
Rate of treatment discontinuation due to toxicity | Through study completion, up until 24 months after the last patient commences treatment
  The percentage of patients who discontinue treatment due to treatment related toxicity will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Arun Azad, Principal Investigator — Peter MacCallum Cancer Centre, Australia; Prof Michael Hofman, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (2):
- Australia (2):
  - St Vincent's Hospital, Sydney, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria